CLINICAL TRIAL: NCT01416441
Title: An Open-Label, Multicenter Study Evaluating the Safety and Tolerability of Once-weekly Oral Aripiprazole in Children and Adolescents With Tourette's Disorder
Brief Title: Safety and Tolerability Study of Once-weekly Oral Aripiprazole in Children and Adolescents With Tourette's Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31-10-274; 2011-000469-11 (EudraCT Number)
Record Dates: First submitted 2011-08-01; First posted 2011-08-15 (Estimated); Results first posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Tourette's Disorder
Keywords: Tourette's Disorder; Tic Disorders
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Aripiprazole (Experimental): Participants received oral aripiprazole tablets once weekly (QW) with a titrated dose starting from 52.5 milligram (mg), on Day 1 and increasing to 77.5 mg and 110 mg for the remainder of the trial (Up to Week 52), the dose could be adjusted between these 3 dose levels as determined by investigator's discretion based on safety and tolerability.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Aripiprazole tablets orally once daily.
  Other Names: ABILIFY

SUMMARY:
The goal of the current trial is to obtain long term efficacy, safety and tolerability data of once weekly aripiprazole in children and adolescents with Tourette's Disorder.

ELIGIBILITY:
Inclusion Criteria:

* The participants successfully completed the final assessment visit in either Study 31-10-272 (NCT01418339) or 31-10-273 (NCT01418352). The participants completed all required assessments for the Week 8/Early Termination Visit to be eligible for rollover in to this open-label trial.
* Written informed consent form (ICF) obtained from a legally acceptable representative & informed assent at Baseline as applicable by trial center's Institutional review board/independent ethics committee (IRB/IEC).
* The participant, designated guardian(s) or caregiver(s) are able to comprehend and satisfactorily comply with the protocol requirements, as evaluated by the investigator.

Exclusion Criteria:

* The participants experienced adverse events (AEs) during the double-blind study 31-10-272 (NCT01418339) or 31-10-273 (NCT01418352) that would, in the investigator's judgment, preclude further exposure to aripiprazole.
* The participants had protocol violations during the double-blind trial considered major in the judgment of the investigator which would deem the participant a poor candidate for the trial.
* A positive drug screen at baseline for cocaine, alcohol or other drugs of abuse which will result in early termination at Week 1.
* Sexually active patients who will not commit to utilizing 2 of the approved birth control methods or who will not remain abstinent during the trial and for 90 and 30 days following the last dose of study drug for male and female respectively.
* Participants representing Risk of committing suicide.
* Body weight lower than 16 kg.
* Abnormal laboratory test results (Platelet, Hemoglobin, Neutrophils, Aspartate aminotransferase, Alanine aminotransferase, Creatinine) vital signs and Electrocardiogram (ECG) results.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 170 (Actual)
Dates: Start 2011-10-19 (Actual); Primary Completion 2014-03-13 (Actual); Study Completion 2014-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Kohegyi, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (72):
- United States (34):
  - Dothan, Alabama
  - Little Rock, Arkansas
  - Los Angeles, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Santa Ana, California
  - Wildomar, California
  - Gainesville, Florida
  - Hialeah, Florida
  - Miami, Florida
  - Orange City, Florida
  - St. Petersburg, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Overland Park, Kansas
  - New Orleans, Louisiana
  - Bloomfield Hills, Michigan
  - Omaha, Nebraska
  - Manhasset, New York
  - Staten Island, New York
  - Avon Lake, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Middleburg Heights, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Bothell, Washington
  - La Crosse, Wisconsin
- Bulgaria (3):
  - Rousse
  - Sofia
  - Varna
- Canada (4):
  - Calgary
  - Kelowna
  - Toronto
  - Whitby
- Germany (5):
  - Aachen
  - Dresden
  - Hanover
  - München
  - Ulm
- Hungary (2):
  - Budapest
  - Szeged
- Mexico (5):
  - Culiacán
  - Durango
  - León
  - Miguel Hidalgo
  - Monterrey
- Romania (4):
  - Bucharest
  - Cluj-Napoca
  - Craiova
  - Iași
- South Korea (4):
  - Gyeonggi-do
  - Gyeongsang
  - Incheon
  - Seoul
- Taiwan (4):
  - Changhua
  - Kaohsiung City
  - Taichung
  - Taipei
- Ukraine (7):
  - Donetsk
  - Kharkiv
  - Kyiv
  - Luhansk
  - Poltava
  - Stepanovka
  - Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/.
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 170 participants were screened and enrolled. 114 participants were enrolled from study 31-10-272 (NCT01418339) and 56 participants were enrolled from study 31-10-273 (NCT01418352). The participants were recruited at 79 sites in following 10 countries: Bulgaria, Canada, Germany, Hungary, Mexico, Romania, South Korea, Taiwan, Ukraine and the US from 19 October 2011 to 13 March 2014.
Pre-assignment Details: Children and adolescents with Tourette's disorder who had successfully completed the previous studies, entered this 52-week open-label extension study to receive once-weekly aripiprazole tablet.
Groups:
- Aripiprazole (Once Weekly): Participants received oral aripiprazole tablets once weekly (QW) with a titrated dose starting from 52.5 milligram (mg), on Day 1 and increasing to 77.5 mg and 110 mg for the remainder of the trial (Up to Week 52), the dose could be adjusted between these 3 dose levels as determined by investigator's discretion based on safety and tolerability.
Period: Overall Study
Arm/Group | Aripiprazole (Once Weekly)
Started | 170
Completed | 89
Not Completed | 81
Not completed — Lost to Follow-up | 5
Not completed — Adverse Event | 6
Not completed — Sponsor Discontinued Trial Site | 43
Not completed — Subject Met Withdrawal Criteria | 10
Not completed — Investigator Withdrew Subject | 2
Not completed — Subject Withdrew Consent | 12
Not completed — Lack of Efficacy as Determined by the Investigator | 3

BASELINE CHARACTERISTICS:
Population: The Enrolled Sample included participants who met the entrance criteria and assigned to the open label treatment (regardless of whether or not they were dosed with study drug).
Arm/Group | Aripiprazole (Once Weekly)
Number analyzed (Participants) | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.2 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31
  Not Hispanic or Latino | 136
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 36
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 117
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  Canada | 19
  South Korea | 15
  Romania | 8
  Hungary | 14
  United States | 50
  Taiwan | 21
  Ukraine | 21
  Mexico | 14
  Bulgaria | 5
  Germany | 3
Weight [Mean (Standard Deviation); unit: Kilogram] | 51.5 (19)
Height [Mean (Standard Deviation); unit: centimeter] | 154.2 (16.4)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilogram per meter square] | 21.0 (4.7)
Time since first diagnosis for Tourette's Disorder [Mean (Standard Deviation); unit: Years] — Time since first diagnosis for Tourette's Disorder (years) = (date of screening assessment - date of first diagnosis + 1)/365.25.
  Years | 2.3 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, Severe TEAEs and TEAEs Leading Treatment Discontinuation
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a participant enrolled in a clinical trial and which did not necessarily have a causal relationship with the study medication. Treatment emergent adverse events (TEAE) are adverse events occurring after the onset of study drug administration.
Time Frame: From signing of the informed consent up to 30 days after the last dose (Up to Week 52)
Population: Safety Sample included all participants who received at least one dose of open-label study medication in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Aripiprazole (Once Weekly)
Number analyzed (Participants) | 170
Participants
  Participants with Serious TEAEs | 5
  Participants with Severe TEAEs | 8
  Participants Discontinued Medication due to TEAE's | 6
  Participants with TEAEs | 104

2. Primary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Parameter Values
Description: The laboratory values were one of the parameters to measure the safety and tolerability of individual participants. Participants with potentially clinically significant lab values in serum chemistry, hematology, urinalyses and prolactin tests that were identified based on pre-defined criteria were reported. Any value outside the normal range was flagged for the attention of the investigator who assessed whether or not a flagged value is of clinical significance.
Time Frame: Baseline to Week 52
Population: Safety Sample included all participants who received at least one dose of open-label study medication in this study. Number analyzed is the number of participants with data available for analyses of the specific category.
Measure: Count of Participants; unit: Participants
Arm/Group | Aripiprazole (Once Weekly)
Number analyzed (Participants) | 170
Participants
  Chemistry-Alkaline Phosphatase: number analyzed (Participants) | 164
  Chemistry-Alkaline Phosphatase | 0
  Chemistry-Alanine Aminotransferase: number analyzed (Participants) | 164
  Chemistry-Alanine Aminotransferase | 1
  Chemistry-Aspartate Aminotransferase: number analyzed (Participants) | 164
  Chemistry-Aspartate Aminotransferase | 1
  Chemistry-Bilirubin, Total: number analyzed (Participants) | 164
  Chemistry-Bilirubin, Total | 4
  Chemistry-Calcium: number analyzed (Participants) | 164
  Chemistry-Calcium | 0
  Chemistry-Chloride: number analyzed (Participants) | 164
  Chemistry-Chloride | 0
  Chemistry-Creatine Phosphokinase: number analyzed (Participants) | 164
  Chemistry-Creatine Phosphokinase | 4
  Chemistry-Creatinine: number analyzed (Participants) | 164
  Chemistry-Creatinine | 0
  Chemistry-Glucose: number analyzed (Participants) | 58
  Chemistry-Glucose | 1
  Chemistry-Glucose, Fasting: number analyzed (Participants) | 146
  Chemistry-Glucose, Fasting | 1
  Chemistry-HDL Cholesterol, Fasting: number analyzed (Participants) | 145
  Chemistry-HDL Cholesterol, Fasting | 3
  Chemistry-Lactic Dehydrogenase: number analyzed (Participants) | 164
  Chemistry-Lactic Dehydrogenase | 1
  Chemistry-LDL-Cholesterol, Fasting: number analyzed (Participants) | 145
  Chemistry-LDL-Cholesterol, Fasting | 2
  Chemistry-Potassium: number analyzed (Participants) | 164
  Chemistry-Potassium | 0
  Chemistry-Sodium: number analyzed (Participants) | 164
  Chemistry-Sodium | 0
  Chemistry- Triglycerides, Fasting: number analyzed (Participants) | 145
  Chemistry- Triglycerides, Fasting | 19
  Chemistry- Urea Nitrogen: number analyzed (Participants) | 164
  Chemistry- Urea Nitrogen | 0
  Chemistry-Uric Acid: number analyzed (Participants) | 164
  Chemistry-Uric Acid | 0
  Urinalysis-Glucose, Urine: number analyzed (Participants) | 156
  Urinalysis-Glucose, Urine | 3
  Urinalysis-Protein, Urine: number analyzed (Participants) | 156
  Urinalysis-Protein, Urine | 1
  Other-Prolactin: number analyzed (Participants) | 159
  Other-Prolactin | 3
  Haematology-Eosinophils: number analyzed (Participants) | 163
  Haematology-Eosinophils | 3
  Haematology-Hematocrit: number analyzed (Participants) | 142
  Haematology-Hematocrit | 0
  Haematology-Hemoglobin: number analyzed (Participants) | 163
  Haematology-Hemoglobin | 3
  Haematology-Neutrophils: number analyzed (Participants) | 163
  Haematology-Neutrophils | 0
  Haematology-Platelet Count: number analyzed (Participants) | 163
  Haematology-Platelet Count | 0
  Haematology-White Blood Count: number analyzed (Participants) | 163
  Haematology-White Blood Count | 4

3. Primary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Values
Description: Incidence of clinically relevant abnormal ECG values were reported as change from Baseline in heart rate (Tachycardia - ≥15 beats per minute (bpm), Bradycardia ≤15 bpm; Rhythm (Sinus tachycardia ≥15 bpm increase, Sinus bradycardia decrease of ≥15 bpm from Baseline); Presence of - supraventricular premature beat; ventricular premature beat; supraventricular tachycardia; ventricular tachycardia; atrial fibrillation and flutter. Conduction - Presence of primary, secondary or tertiary atrioventricular block, left bundle-branch block, right bundle-branch block, pre-excitation syndrome, other intraventricular conduction blocked QRS ≥0.12 second increase of ≥0.02 second. Acute, subacute or old Infarction, Presence of myocardial ischemia, symmetrical T-wave inversion. Increase in QTc - QTc ≥450 msec ≥10% increase. Any clinically significant change from Baseline assessed by the Investigator are reported.
Time Frame: Baseline to Week 52
Population: Safety Sample included all participants who received at least one dose of open-label study medication in this study, with data available for analyses.
Measure: Number; unit: participants
Arm/Group | Aripiprazole (Once Weekly)
Number analyzed (Participants) | 154
participants
  Tachycardia | 1
  Bradycardia | 0
  Sinus Tachycardia | 1
  Sinus Bradycardia | 0
  Supraventricular Premature Beat | 4
  Ventricular Premature Beat | 3
  Supraventricular Tachycardia | 0
  Ventricular Tachycardia | 0
  Atrial Fibrillation | 0
  Atrial Flutter | 0
  Primary Atrioventricular Block | 0
  Secondary Atrioventricular Block | 0
  Tertiary Atrioventricular Block | 0
  Left Bundle Branch Block | 0
  Right Bundle Branch Block | 2
  Pre-excitation Syndrome | 0
  Other intraventricular conduction block | 0
  Acute or Sub-acute Infarction | 0
  Old Infarction | 0
  Myocardial Ischemia | 0
  Symmetrical T-Wave Inversion | 1
  QT Interval cCorrected for Heart Rate by Bazett's Formula (QTB) | 3
  QT Interval Corrected for Heart Rate by Fredericia's Formula (QTcF) | 0
  QT Interval Corrected for Heart Rate by the US Food and Drug (QTcN) | 1

4. Primary Outcome: Number of Participants With Emergence of Suicidal Ideation, TEAEs Related to Suicide and Suicidality and Suicide Ideation From the Potential Suicide Events Recorded on the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: Suicidality was defined as reporting at least one occurrence of any suicidal behavior or suicidal ideation. Suicidal behavior was defined as reporting any type of suicidal behaviors (actual attempt, interrupted attempt, aborted attempt, and preparatory acts or behavior). Suicidal ideation was defined as reporting any type of suicidal ideation. The suicidal ideation intensity total score is the sum of intensity scores of 5 items (frequency, duration, controllability, deterrents, and reasons for ideation). The score of each intensity item ranges from 0 (none) to 5 (worst) which leads to the range of the total score from 0 to 25. A missing score of any item resulted in a missing total score. If no suicidal ideation was reported, a score of 0 was given to the intensity scale.
Time Frame: Baseline to Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Aripiprazole (Once Weekly)
Number analyzed (Participants) | 170
Participants
  Emergence of Suicidal Ideation: number analyzed (Participants) | 167
  Emergence of Suicidal Ideation | 3
  TEAEs related to Suicide | 3
  Suicidality and Suicidal Ideation: number analyzed (Participants) | 169
  Suicidality and Suicidal Ideation | 4

5. Primary Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Score
Description: The AIMS Scale is an extrapyramidal symptoms (EPS) rating scale. The AIMS is a 12 item scale. The first 10 items e.g. facial and oral movements (items 1-4), extremity movements (items 5 and 6), trunk movements (item 7), investigators global assessment of dyskinesia (items 8 to 10) are rated from 0 to 4 (0=best, 4=worst). Items 11 and 12, related to dental status, have dichotomous responses, 0=no and 1=yes. The AIMS Total Score is the sum of the ratings for the first seven items. The possible total scores are from 0 to 28. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 32, 40, 52; Last Visit (Week 52 or early termination Visit before Week 52)
Population: Safety Sample included all participants who received at least one dose of open-label study medication in this study. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aripiprazole (Once Weekly)
Number analyzed (Participants) | 170
score on a scale
  Change at Week 4: number analyzed (Participants) | 163
  Change at Week 4 | -0.1 (1.3)
  Change at Week 8: number analyzed (Participants) | 158
  Change at Week 8 | -0.1 (1.6)
  Change at Week 12: number analyzed (Participants) | 152
  Change at Week 12 | -0.4 (1.7)
  Change at Week 16: number analyzed (Participants) | 147
  Change at Week 16 | -0.5 (2)
  Change at Week 20: number analyzed (Participants) | 134
  Change at Week 20 | -0.5 (2)
  Change at Week 24: number analyzed (Participants) | 123
  Change at Week 24 | -0.6 (2.5)
  Change at Week 32: number analyzed (Participants) | 114
  Change at Week 32 | -0.8 (2.3)
  Change at Week 40: number analyzed (Participants) | 104
  Change at Week 40 | -0.8 (2.4)
  Change at Week 52: number analyzed (Participants) | 90
  Change at Week 52 | -0.9 (2.4)
  Change at Last Visit (Early Termination Visit Prior to or at Week 52: number analyzed (Participants) | 168
  Change at Last Visit (Early Termination Visit Prior to or at Week 52 | -0.8 (2.3)

6. Primary Outcome: Mean Change From Baseline in Body Mass Index (BMI)
Description: The BMI kilogram/meter square (i.e. kg/m^2) was calculated from the Baseline height and the weight at the current visit using one of the following formulae, as appropriate: Weight (kg) divided by [Height (meters)]^2.
Time Frame: Baseline and Weeks 12, 24, 52 and Last Visit (Week 52 or early termination Visit before Week 52)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Aripiprazole (Once Weekly)
Number analyzed (Participants) | 170
kg/m^2
  Change at Week 12: number analyzed (Participants) | 150
  Change at Week 12 | 0.6 (0.9)
  Change at Week 24: number analyzed (Participants) | 122
  Change at Week 24 | 0.4 (1.5)
  Change at Week 52: number analyzed (Participants) | 90
  Change at Week 52 | 0.7 (2)
  Change at Last Visit (Early Termination Visit Prior to or at Week 52: number analyzed (Participants) | 166
  Change at Last Visit (Early Termination Visit Prior to or at Week 52 | 0.6 (1.8)

7. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital signs assessments included orthostatic (supine and standing) blood pressure (BP) measured as millimeter of mercury [mmHg]), heart rate, (measured in beats per minute [bpm]), body weight (measured in kilograms [kg]) and body temperature. Incidence of clinically relevant abnormal values in heart rate, systolic and diastolic blood pressure and weight were identified based on pre-defined criteria. Orthostatic assessments of blood pressure and heart rate were made after the participant has been supine for at least 5 minutes and again after the participant has been standing for approximately 2 minutes, but not more than 3 minutes.
Time Frame: Baseline to Week 52
Population: Safety Sample included all participants who received at least one dose of open-label study medication in this study. Number analyzed is the number of participants with data available for analyses of the specific category at given timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Aripiprazole (Once Weekly)
Number analyzed (Participants) | 170
Participants
  Heart Rate Supine- Increase ≥15 bpm: number analyzed (Participants) | 168
  Heart Rate Supine- Increase ≥15 bpm | 1
  Heart Rate Supine- Decrease ≥15 bpm: number analyzed (Participants) | 168
  Heart Rate Supine- Decrease ≥15 bpm | 0
  Heart Rate Standing-increase ≥15 bpm: number analyzed (Participants) | 167
  Heart Rate Standing-increase ≥15 bpm | 4
  Heart Rate Standing- Decrease ≥15 bpm: number analyzed (Participants) | 167
  Heart Rate Standing- Decrease ≥15 bpm | 0
  Systolic Supine BP- Increase ≥20 mmHg: number analyzed (Participants) | 168
  Systolic Supine BP- Increase ≥20 mmHg | 0
  Systolic Supine BP- Decrease ≥20 mmHg: number analyzed (Participants) | 168
  Systolic Supine BP- Decrease ≥20 mmHg | 1
  Systolic Standing BP- Increase ≥20 mmHg: number analyzed (Participants) | 167
  Systolic Standing BP- Increase ≥20 mmHg | 0
  Systolic Standing BP- Decrease ≥20 mmHg: number analyzed (Participants) | 167
  Systolic Standing BP- Decrease ≥20 mmHg | 1
  Diastolic Supine BP- Increase ≥15 mmHg: number analyzed (Participants) | 168
  Diastolic Supine BP- Increase ≥15 mmHg | 0
  Diastolic Supine BP- Decrease ≥15 mmHg: number analyzed (Participants) | 168
  Diastolic Supine BP- Decrease ≥15 mmHg | 0
  Diastolic Standing BP- Increase ≥15 mmHg: number analyzed (Participants) | 167
  Diastolic Standing BP- Increase ≥15 mmHg | 1
  Diastolic Standing BP- Decrease ≥15 mmHg: number analyzed (Participants) | 167
  Diastolic Standing BP- Decrease ≥15 mmHg | 0
  Orthostatic Hypotension: number analyzed (Participants) | 169
  Orthostatic Hypotension | 2
  Weight-Gain ≥ 7%: number analyzed (Participants) | 166
  Weight-Gain ≥ 7% | 82
  Weight-Loss ≥ 7%: number analyzed (Participants) | 166
  Weight-Loss ≥ 7% | 6

8. Primary Outcome: Mean Change From Baseline in Simpson Angus Scale (SAS) Score
Description: The SAS is a rating scale used to measure Extrapyramidal symptoms (EPS). The SAS scale consists of a list of 10 symptoms of parkinsonism (gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, head rotation, glabella tap, tremor, salivation, and akathisia), with each item rated from 0 to 4, with 0 being normal and 4 being the worst. The SAS Total score is sum of ratings for all 10 items, with possible Total scores from 0 to 40. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 32, 40, 52; Last Visit (Week 52 or early termination Visit before Week 52)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Aripiprazole (Once Weekly)
Number analyzed (Participants) | 170
score on scale
  Change at Week 4: number analyzed (Participants) | 163
  Change at Week 4 | 0 (0.3)
  Change at Week 8: number analyzed (Participants) | 158
  Change at Week 8 | 0 (0.4)
  Change at Week 12: number analyzed (Participants) | 152
  Change at Week 12 | 0 (0.3)
  Change at Week 16: number analyzed (Participants) | 147
  Change at Week 16 | 0 (0.4)
  Change at Week 20: number analyzed (Participants) | 134
  Change at Week 20 | 0 (0.2)
  Change at Week 24: number analyzed (Participants) | 123
  Change at Week 24 | 0 (0.5)
  Change at Week 32: number analyzed (Participants) | 114
  Change at Week 32 | 0 (0.4)
  Change at Week 40: number analyzed (Participants) | 104
  Change at Week 40 | 0 (0.5)
  Change at Week 52: number analyzed (Participants) | 89
  Change at Week 52 | 0 (0.5)
  Change at Last Visit (Week 52 or early termination Visit before Week 52): number analyzed (Participants) | 168
  Change at Last Visit (Week 52 or early termination Visit before Week 52) | 0 (0.4)

9. Primary Outcome: Mean Change From Baseline in Barnes Akathisia Rating Scale (BARS) Score
Description: The BARS was an EPS rating scale. The BARS was used to assess the presence and severity of akathisia. This scale consists of 4 items. Only the 4th item, the Global Clinical Assessment of Akathisia, was evaluated in this trial. This item is rated on a 6 point scale, with 0 being best (absent) and 5 being worst (severe akathisia). A negative change from Baseline indicates improvement.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 32,40, 52; Last Visit (Week 52 or early termination Visit before Week 52)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aripiprazole (Once Weekly)
Number analyzed (Participants) | 170
score on a scale
  Change at Week 4: number analyzed (Participants) | 163
  Change at Week 4 | 0 (0.3)
  Change at Week 8: number analyzed (Participants) | 158
  Change at Week 8 | 0 (0.2)
  Change at Week 12: number analyzed (Participants) | 152
  Change at Week 12 | 0 (0.2)
  Change at Week 16: number analyzed (Participants) | 147
  Change at Week 16 | 0 (0.2)
  Change at Week 20: number analyzed (Participants) | 134
  Change at Week 20 | 0 (0.2)
  Change at Week 24: number analyzed (Participants) | 123
  Change at Week 24 | 0 (0.1)
  Change at Week 32: number analyzed (Participants) | 114
  Change at Week 32 | 0 (0.2)
  Change at Week 40: number analyzed (Participants) | 104
  Change at Week 40 | 0 (0.2)
  Change at Week 52: number analyzed (Participants) | 90
  Change at Week 52 | 0 (0.3)
  Change at Last Visit (Week 52 or early termination Visit before Week 52): number analyzed (Participants) | 168
  Change at Last Visit (Week 52 or early termination Visit before Week 52) | 0 (0.3)

10. Primary Outcome: Mean Change From Baseline in Average Score of Attention-Deficit Disorder/Attention-Deficit Hyperactivity Disorder (ADD/ADHD) Sub-scale of the Swanson, Nolan and Pelham-IV (SNAP-IV)
Description: The SNAP-IV, ADHD Inattention subscale contains 19 items, items 1 to 9 measure inattention, items 11 to 19 measure hyperactivity/impulsivity, and item 10 for inattention domain that scores the intensity of each item during the last seven days on a 0 to 3 scale (0=not at all, 1=just a little, 2=pretty much, 3=very much). The lowest possible score is 0; highest is 57. The negative change from Baseline indicates improvement.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 32,40, 52; Last Visit (Week 52 or early termination Visit before Week 52)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aripiprazole (Once Weekly)
Number analyzed (Participants) | 170
score on a scale
  Change at Week 4: number analyzed (Participants) | 163
  Change at Week 4 | -0.1 (0.3)
  Change at Week 8: number analyzed (Participants) | 158
  Change at Week 8 | 0 (0.3)
  Change at Week 12: number analyzed (Participants) | 152
  Change at Week 12 | -0.1 (0.3)
  Change at Week 16: number analyzed (Participants) | 147
  Change at Week 16 | -0.1 (0.4)
  Change at Week 20: number analyzed (Participants) | 134
  Change at Week 20 | -0.1 (0.3)
  Change at Week 24: number analyzed (Participants) | 123
  Change at Week 24 | -0.2 (0.4)
  Change at Week 32: number analyzed (Participants) | 114
  Change at Week 32 | -0.2 (0.4)
  Change at Week 40: number analyzed (Participants) | 104
  Change at Week 40 | -0.2 (0.4)
  Change at Week 52: number analyzed (Participants) | 90
  Change at Week 52 | -0.1 (0.4)
  Change at Last Visit (Week 52 or early termination Visit before Week 52): number analyzed (Participants) | 168
  Change at Last Visit (Week 52 or early termination Visit before Week 52) | -0.1 (0.4)

11. Primary Outcome: Mean Change From Baseline in Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) Total Score
Description: The CY-BOCS is used to assess characteristics of obsession and compulsion for the week prior to the interview. Nineteen items are rated in the CY-BOCS, but the total score is the sum of only items 1 to 10 (excluding items 1b and 6b). The obsession and compulsion subtotals are the sums of items 1 to 5 (excluding 1b) and 6 to 10 (excluding 6b), respectively. A missing value for any CY-BOCS item scale could result in a missing total score or obsession and compulsion subtotals of which the item scale is a component. At baseline, the full CY-BOCS interview is conducted. At all post-baseline time points, the "Questions on Obsessions" (items 1 to 5) and "Questions on Compulsions" (items 6 to 10) are reviewed and the target symptoms identified at baseline are the primary focus for rating severity. CY-BOCS total score could range from 0 to 40. Higher scores indicate worse outcome. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 32,40, 52; Last Visit (Week 52 or early termination Visit before Week 52)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aripiprazole (Once Weekly)
Number analyzed (Participants) | 170
score on a scale
  Change at Week 4: number analyzed (Participants) | 163
  Change at Week 4 | -0.2 (1.6)
  Change at Week 8: number analyzed (Participants) | 158
  Change at Week 8 | -0.2 (1.9)
  Change at Week 12: number analyzed (Participants) | 152
  Change at Week 12 | -0.3 (1.8)
  Change at Week 16: number analyzed (Participants) | 147
  Change at Week 16 | -0.4 (1.9)
  Change at Week 20: number analyzed (Participants) | 134
  Change at Week 20 | -0.4 (2)
  Change at Week 24: number analyzed (Participants) | 123
  Change at Week 24 | -0.5 (2.2)
  Change at Week 32: number analyzed (Participants) | 114
  Change at Week 32 | -0.6 (2.5)
  Change at Week 40: number analyzed (Participants) | 104
  Change at Week 40 | -0.6 (2.4)
  Change at Week 52: number analyzed (Participants) | 90
  Change at Week 52 | -0.3 (2.4)
  Change at Last Visit (Week 52 or early termination Visit before Week 52): number analyzed (Participants) | 168
  Change at Last Visit (Week 52 or early termination Visit before Week 52) | -0.3 (2.4)

12. Primary Outcome: Mean Change From Baseline in Children's Depression Rating Scale Revised (CDRS-R) Total Score
Description: The CDRS-R is composed of 17 interviewer-rated symptom areas: impaired schoolwork, difficulty having fun, social withdrawal, appetite disturbance, sleep disturbance, excessive fatigue, physical complaints, irritability, excessive guilt, low self-esteem, depressed feelings, morbid ideas, suicidal ideas, excessive weeping, depressed facial affect, listless speech, and hypoactivity. The CDRS-R total score is the sum of scores for the 17 symptom areas. A missing value for any CDRS-R item scale or a not rated item scale (indicated by the value of 0) could result in a missing total score. The CDRS-R total score is the sum of scores for the 17 symptom areas and could range from 17 to 113 with higher values indicating worse outcome. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 32,40, 52; Last Visit (Week 52 or early termination Visit before Week 52)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aripiprazole (Once Weekly)
Number analyzed (Participants) | 170
score on a scale
  Change at Week 4: number analyzed (Participants) | 163
  Change at Week 4 | 0 (2.3)
  Change at Week 8: number analyzed (Participants) | 158
  Change at Week 8 | 0 (2.6)
  Change at Week 12: number analyzed (Participants) | 152
  Change at Week 12 | -0.2 (3.1)
  Change at Week 16: number analyzed (Participants) | 147
  Change at Week 16 | -0.4 (2.9)
  Change at Week 20: number analyzed (Participants) | 134
  Change at Week 20 | -0.3 (3.1)
  Change at Week 24: number analyzed (Participants) | 123
  Change at Week 24 | -0.2 (2.5)
  Change at Week 32: number analyzed (Participants) | 114
  Change at Week 32 | -0.1 (2.8)
  Change at Week 40: number analyzed (Participants) | 104
  Change at Week 40 | -0.4 (2.7)
  Change at Week 52: number analyzed (Participants) | 90
  Change at Week 52 | -0.2 (3.3)
  Change at Last Visit (Week 52 or early termination Visit before Week 52): number analyzed (Participants) | 168
  Change at Last Visit (Week 52 or early termination Visit before Week 52) | 0.3 (4.1)

13. Primary Outcome: Mean Change From Baseline in Pediatric Anxiety Rating Scale (PARS) Total Severity Score
Description: The PARS has 2 sections: the symptom checklist and the severity items. The symptom checklist is used to determine the child's repertoire of symptoms during the past week. Information is elicited from the child and parent(s) and the rater then combines information from all informants using his/her best judgment. The 7-item severity list is used to determine severity of symptoms and the PARS total score. The time frame for the PARS rating is the past week. Only those symptoms endorsed for the past week are included in the symptom checklist and rated on the severity items. The PARS total severity score is the sum of items 2, 3, 5, 6, and 7. The total severity score ranges from 0 to 25, with 25 being the worst. Codes "8" (Not applicable) and "9" (Does not know) are not included in the summation (ie, equivalent to a score of 0 in the summation). A negative change from Baseline indicates improvement.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 32,40, 52; Last Visit (Week 52 or early termination Visit before Week 52)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aripiprazole (Once Weekly)
Number analyzed (Participants) | 170
score on a scale
  Change at Week 4: number analyzed (Participants) | 165
  Change at Week 4 | -0.1 (2.6)
  Change at Week 8: number analyzed (Participants) | 158
  Change at Week 8 | -0.2 (2.4)
  Change at Week 12: number analyzed (Participants) | 152
  Change at Week 12 | -0.3 (1.8)
  Change at Week 16: number analyzed (Participants) | 151
  Change at Week 16 | -0.3 (2)
  Change at Week 20: number analyzed (Participants) | 134
  Change at Week 20 | -0.3 (2.1)
  Change at Week 24: number analyzed (Participants) | 125
  Change at Week 24 | -0.3 (2.3)
  Change at Week 32: number analyzed (Participants) | 116
  Change at Week 32 | -0.3 (2.4)
  Change at Week 40: number analyzed (Participants) | 111
  Change at Week 40 | -0.6 (2.3)
  Change at Week 52: number analyzed (Participants) | 90
  Change at Week 52 | -0.7 (2.4)
  Change at Last Visit (Week 52 or early termination Visit before Week 52): number analyzed (Participants) | 168
  Change at Last Visit (Week 52 or early termination Visit before Week 52) | -0.3 (2.6)

14. Primary Outcome: Mean Change From Baseline in Body Weight
Time Frame: Baseline to Weeks 12, 24, 52 and Last Visit (Week 52 or early termination Visit before Week 52)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Aripiprazole (Once Weekly)
Number analyzed (Participants) | 170
kilogram
  Change at Week 12: number analyzed (Participants) | 151
  Change at Week 12 | 1.4 (2.3)
  Change at Week 24: number analyzed (Participants) | 123
  Change at Week 24 | 2.5 (3.9)
  Change at Week 52: number analyzed (Participants) | 90
  Change at Week 52 | 4.7 (6)
  Change at Last Visit (Week 52 or early termination Visit before Week 52): number analyzed (Participants) | 166
  Change at Last Visit (Week 52 or early termination Visit before Week 52) | 3.8 (5.1)

15. Primary Outcome: Mean Change From Baseline in Waist Circumference
Description: Waist circumference was recorded before a participant's meal and at approximately the same time at each visit. Measurement was accomplished by locating the upper hip bone and the top of the right iliac crest and placing the measuring tape in a horizontal plane around the abdomen at the level of the crest. Before reading the tape measure, the assessor assured that the tape was snug, but did not compress the skin, and is parallel to the floor. The measurement was made at the end of a normal exhalation.
Time Frame: Baseline to Weeks 12, 24, 52 and Last Visit (Week 52 or early termination Visit before Week 52)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Aripiprazole (Once Weekly)
Number analyzed (Participants) | 170
centimeter
  Change at Week 12: number analyzed (Participants) | 150
  Change at Week 12 | 0.4 (3.9)
  Change at Week 24: number analyzed (Participants) | 122
  Change at Week 24 | 1 (5.2)
  Change at Week 52: number analyzed (Participants) | 90
  Change at Week 52 | 2.3 (6.8)
  Change at Last Visit (Week 52 or early termination Visit before Week 52): number analyzed (Participants) | 166
  Change at Last Visit (Week 52 or early termination Visit before Week 52) | 1.9 (5.8)

16. Secondary Outcome: Mean Change From Baseline in Yale Global Tic Severity Scale (YGTSS) Total Tic Score
Description: The YGTSS is a semi-structured clinical interview designed to measure the tic severity. This scale consisted of a tic inventory, with 5 separate rating scales to rate the severity of symptoms, and an impairment ranking. Ratings were made along 5 different dimensions on a scale of 0 to 5 for motor and vocal tics, each including number, frequency, intensity, complexity, and interference. The YGTSS TTS was the summation of the severity scores of motor and vocal tics. The total tic score (TTS) ranged from 0 (none) to 50 (severe) with higher score represent more severe symptoms (A negative change from Baseline indicates improvement).
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 32,40, 52; Last Visit (Week 52 or early termination Visit before Week 52)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Aripiprazole (Once Weekly)
Number analyzed (Participants) | 170
score on scale
  Change at Week 4: number analyzed (Participants) | 163
  Change at Week 4 | -2.6 (5.4)
  Change at Week 8: number analyzed (Participants) | 158
  Change at Week 8 | -3.8 (5.6)
  Change at Week 12: number analyzed (Participants) | 152
  Change at Week 12 | -4.5 (6.7)
  Change at Week 16: number analyzed (Participants) | 147
  Change at Week 16 | -4.6 (6.8)
  Change at Week 20: number analyzed (Participants) | 134
  Change at Week 20 | -5.5 (7.2)
  Change at Week 24: number analyzed (Participants) | 123
  Change at Week 24 | -5.8 (7.9)
  Change at Week 32: number analyzed (Participants) | 114
  Change at Week 32 | -6 (9.1)
  Change at Week 40: number analyzed (Participants) | 104
  Change at Week 40 | -6.4 (9.3)
  Change at Week 52: number analyzed (Participants) | 90
  Change at Week 52 | -5.8 (8.8)
  Change at Last Visit (Week 52 or early termination Visit before Week 52): number analyzed (Participants) | 168
  Change at Last Visit (Week 52 or early termination Visit before Week 52) | -5.9 (8.4)

17. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression for Tourette's Syndrome (CGI-TS) Severity of Illness Score
Description: The severity of illness and efficacy of study medication for each participant were rated using the CGI-TS scale. The study physician rated the participants total improvement whether or not it is due to study treatment. All responses were compared to the participants condition at Baseline (Day 0). Response choices include: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 32,40, 52; Last Visit (Week 52 or early termination Visit before Week 52)
Population: Efficacy Sample included all participants who received at least one dose of open-label study medication in this study and had a baseline and at least one post baseline efficacy evaluation. Number analyzed is the number of participants with data available for the analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aripiprazole (Once Weekly)
Number analyzed (Participants) | 170
score on a scale
  Change at Week 4: number analyzed (Participants) | 163
  Change at Week 4 | -0.2 (0.7)
  Change at Week 8: number analyzed (Participants) | 158
  Change at Week 8 | -0.4 (0.8)
  Change at Week 12: number analyzed (Participants) | 152
  Change at Week 12 | -0.4 (0.8)
  Change at Week 16: number analyzed (Participants) | 147
  Change at Week 16 | -0.5 (0.8)
  Change at Week 20: number analyzed (Participants) | 134
  Change at Week 20 | -0.6 (0.8)
  Change at Week 24: number analyzed (Participants) | 123
  Change at Week 24 | -0.5 (0.9)
  Change at Week 32: number analyzed (Participants) | 114
  Change at Week 32 | -0.6 (1)
  Change at Week 40: number analyzed (Participants) | 104
  Change at Week 40 | -0.7 (1.1)
  Change at Week 52: number analyzed (Participants) | 90
  Change at Week 52 | -0.7 (1.1)
  Change at Last Visit (Week 52 or early termination Visit before Week 52): number analyzed (Participants) | 168
  Change at Last Visit (Week 52 or early termination Visit before Week 52) | -0.6 (1.1)

18. Secondary Outcome: Mean Change From Baseline in Total YGTSS Score
Description: The YGTSS consists of a tic inventory, with 5 separate rating scales to rate the severity of symptoms (on a scale of 0 to 5 for 5 different dimensions, including number, frequency, intensity, complexity, and interference) of motor and vocal tics, and an impairment ranking. The Total YGTSS score is the summation of the severity scores of motor and vocal tics and also the ranking of impairment (range of 0 to 100). A missing value of a YGTSS item scale could result in a missing Total YGTSS score. A negative change in Total YGTSS score from baseline represents an improvement in symptoms.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 32,40, 52; Last Visit (Week 52 or early termination Visit before Week 52)
Population: Safety Sample included all participants who received at least one dose of open-label study medication in this study. Number analyzed is the number of participants with data available for the analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aripiprazole (Once Weekly)
Number analyzed (Participants) | 170
score on a scale
  Change at Week 4: number analyzed (Participants) | 163
  Change at Week 4 | -5.6 (10.4)
  Change at Week 8: number analyzed (Participants) | 158
  Change at Week 8 | -7.4 (11.8)
  Change at Week 12: number analyzed (Participants) | 152
  Change at Week 12 | -8.6 (12.9)
  Change at Week 16: number analyzed (Participants) | 147
  Change at Week 16 | -9.4 (13.9)
  Change at Week 20: number analyzed (Participants) | 134
  Change at Week 20 | -10.7 (14.9)
  Change at Week 24: number analyzed (Participants) | 123
  Change at Week 24 | -10.4 (16)
  Change at Week 32: number analyzed (Participants) | 114
  Change at Week 32 | -11.6 (17.5)
  Change at Week 40: number analyzed (Participants) | 104
  Change at Week 40 | -12.6 (17.5)
  Change at Week 52: number analyzed (Participants) | 90
  Change at Week 52 | -10.8 (17.4)
  Change at Last Visit (Week 52 or early termination Visit before Week 52): number analyzed (Participants) | 168
  Change at Last Visit (Week 52 or early termination Visit before Week 52) | -11.4 (16.7)

19. Secondary Outcome: Response Rates
Description: Response rates - clinical response was defined as percentage of participants >25% improvement from Baseline to endpoint in YGTSS TTS OR a CGI-TS change score of 1 [very much improved] or 2 [much improved] at endpoint. The YGTSS consists of a tic inventory, with 5 separate rating scales to rate the severity of symptoms (on a scale of 0 to 5 for 5 different dimensions, including number, frequency, intensity, complexity, and interference) of motor and vocal tics, and an impairment ranking. The Total YGTSS score is the summation of the severity scores of motor and vocal tics and also the ranking of impairment (range of 0 to 100) with higher score representing severe symptoms.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 32,40, 52; Last Visit (Week 52 or early termination Visit before Week 52)
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | Aripiprazole (Once Weekly)
Number analyzed (Participants) | 170
percentage of participants
  Week 4: number analyzed (Participants) | 163
  Week 4 | 66.2
  Week 8: number analyzed (Participants) | 158
  Week 8 | 69.7
  Week 12: number analyzed (Participants) | 152
  Week 12 | 72.6
  Week 16: number analyzed (Participants) | 147
  Week 16 | 72.3
  Week 20: number analyzed (Participants) | 134
  Week 20 | 74.2
  Week 24: number analyzed (Participants) | 123
  Week 24 | 71.8
  Week 32: number analyzed (Participants) | 114
  Week 32 | 77.8
  Week 40: number analyzed (Participants) | 104
  Week 40 | 80.8
  Week 52: number analyzed (Participants) | 90
  Week 52 | 76.5
  Last Visit (Week 52 or early termination Visit before Week 52) | 71.3

20. Secondary Outcome: Treatment Discontinuation Rates
Description: Treatment discontinuation rate was calculated as the percentage of participants who discontinued treatment.
Time Frame: Up to Week 53
Population: Enrolled Sample include all participants who met the entrance criteria and enrolled in the trial.
Measure: Number; unit: percentage of participants
Arm/Group | Aripiprazole (Once Weekly)
Number analyzed (Participants) | 170
percentage of participants
  All reasons | 47.6
  Other than sponsor discontinued study site | 22.4

21. Secondary Outcome: Mean Change From Baseline in Gilles de la Tourette Quality of Life (GTS-QOL) Overall Score
Description: The GTS-QOL is a disease-specific patient-reported scale for the measurement of health-related quality of life in participants with Tourette's Disorder, taking into account the complexity of the clinical picture of the disease. The questionnaire consists of a 27-item Tourette's Disorder-specific scale with 4 subscales (psychological, physical, obsessional, and cognitive). The GTS-QOL total score ranged from 0 (extremely dissatisfied with life) and 100 (extremely satisfied with life). A positive change from Baseline indicates improvement.
Time Frame: Baseline and Weeks 4, 24, 52 and Last Visit (Week 52 or early termination Visit before Week 52)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aripiprazole (Once Weekly)
Number analyzed (Participants) | 170
score on a scale
  Change at Week 4: number analyzed (Participants) | 168
  Change at Week 4 | -2.9 (8.2)
  Change at Week 24: number analyzed (Participants) | 123
  Change at Week 24 | -3.6 (11.3)
  Change at Week 52: number analyzed (Participants) | 89
  Change at Week 52 | -4.3 (10.5)
  Change at Last Visit (Week 52 or early termination Visit before Week 52): number analyzed (Participants) | 168
  Change at Last Visit (Week 52 or early termination Visit before Week 52) | -3.8 (10.9)

ADVERSE EVENTS:
Time Frame: From first dose up to 4 weeks post last dose (Up to 56 weeks)
Arm/Group | Aripiprazole (Once Weekly)
All-Cause Mortality (participants affected / at risk) | 0/170
Serious Adverse Events (participants affected / at risk) | 5/170
Other Adverse Events (participants affected / at risk) | 57/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole (Once Weekly) (N=170)
Blood creatinine phosphokinase increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Tourette's disorder (Congenital, familial and genetic disorders) | 1
Tremor (Nervous system disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1
Appendicitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole (Once Weekly) (N=170)
Weight increased (Investigations) | 14
Headache (Nervous system disorders) | 19
Somnolence (Nervous system disorders) | 11
Nausea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 12
Nasopharyngitis (Infections and infestations) | 12
Upper respiratory tract infection (Infections and infestations) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.